CLINICAL TRIAL: NCT00933231
Title: A Comparison of Effects of Standard Dose vs. Low Dose Advagraf® With IL-2 Receptor Antibody Induction, MMF and Steroids, With or Without ACEi/ARB - Based Antihypertensive Therapy on Renal Allograft Histology, Function, and Immune Response
Brief Title: Comparison of Standard Versus Low Dose Advagraf® With or Without Angiotensin-converting Enzyme Inhibitor (ACEi)/Angiotensin Receptor Blocker (ARB) on Histology and Function of Renal Allografts
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma Canada, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: FKC-014
Record Dates: First submitted 2009-07-02; First posted 2009-07-07 (Estimated); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Kidney Transplantation
Keywords: Tacrolimus; Kidney Transplantation; Advagraf; Immunosuppression; Angiotensin-Converting Enzyme Inhibitors
MeSH Terms: interventions — Tacrolimus; Basiliximab; Mycophenolic Acid; Adrenal Cortex Hormones; Methylprednisolone; Prednisone; Ramipril; Irbesartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Tacrolimus Standard Dose with ACEi/ARB (Active Comparator): Participants receive a standard dose of tacrolimus with ACEi/ARB.
  Interventions: Drug: tacrolimus; Biological: Simulect; Drug: Cellcept; Drug: Corticosteroids; Drug: Ramipril; Drug: Irbesartan
- Tacrolimus Standard Dose without ACEi/ARB (Active Comparator): Participants receive a standard dose of tacrolimus without ACEi/ARB.
  Interventions: Drug: tacrolimus; Biological: Simulect; Drug: Cellcept; Drug: Corticosteroids
- Tacrolimus Low Dose with ACEi/ARB (Experimental): Participants receive a low dose of tacrolimus with ACEi/ARB.
  Interventions: Drug: tacrolimus; Biological: Simulect; Drug: Cellcept; Drug: Corticosteroids; Drug: Ramipril; Drug: Irbesartan
- Tacrolimus Low Dose without ACEi/ARB (Experimental): Participants receive a low dose of tacrolimus without ACEi/ARB.
  Interventions: Drug: tacrolimus; Biological: Simulect; Drug: Cellcept; Drug: Corticosteroids

INTERVENTIONS:
Drug: tacrolimus — Standard dose, Oral
  Other Names: Advagraf; FK506XL; Prolonged Release Tacrolimus; Tacrolimus XL; Extended Release Tacrolimus; FK506E; MR4
  Arms: Tacrolimus Standard Dose with ACEi/ARB; Tacrolimus Standard Dose without ACEi/ARB
Drug: tacrolimus — Low dose, Oral
  Other Names: Prolonged Release Tacrolimus; FK506XL; Extended Release Tacrolimus; Tacrolimus XL; FK506E; MR4; Advagraf
  Arms: Tacrolimus Low Dose with ACEi/ARB; Tacrolimus Low Dose without ACEi/ARB
Biological: Simulect — IV
  Other Names: Basiliximab
Drug: Cellcept — Oral
  Other Names: MMF
Drug: Corticosteroids — IV and Oral
  Other Names: Methylprednisolone; prednisone
Drug: Ramipril — Oral
  Other Names: Altace; ACEi
  Arms: Tacrolimus Low Dose with ACEi/ARB; Tacrolimus Standard Dose with ACEi/ARB
Drug: Irbesartan — Oral
  Other Names: Avapro; ARB
  Arms: Tacrolimus Low Dose with ACEi/ARB; Tacrolimus Standard Dose with ACEi/ARB

SUMMARY:
This is a multicentre study examining the use of Advagraf-minimization strategy and/or the use of an inhibitor of the renin-angiotensin system in reducing chronic rejection in renal allografts.

DETAILED DESCRIPTION:
The study will consist of the following 4 treatment groups.:

1. Standard dose Advagraf with angiotensin-converting enzyme inhibitor (ACEi)/angiotensin receptor blocker (ARB) antihypertensive therapy
2. Standard dose Advagraf without ACEi/ARB antihypertensive therapy
3. Low dose Advagraf with ACEi/ARB antihypertensive therapy
4. Low dose Advagraf without ACEi/ARB antihypertensive therapy

ELIGIBILITY:
Inclusion Criteria:

* Subject is the recipient of a first or second deceased or living donor renal transplant (one kidney only)
* Subject must have at least one HLA-mismatch with the donor. HLA identical donor-recipient pairs are not eligible
* Subject understands either English or French
* If female and of child-bearing potential, subject has a negative pregnancy test and utilizes adequate contraceptive methods

Exclusion Criteria:

* Presence of donor specific antibody
* Subject who is currently participating in a study with investigational drug, or who has received investigational drug within three months prior to randomization. Observational studies are acceptable
* Subject who has lost a previous graft for immunological reasons less than one year from transplant
* Subject is pregnant or breastfeeding
* Subject receives a kidney lacking pre-implantation biopsy
* Subject has significant disease (e.g. malignancy or uncontrolled infection) or disability (e.g. cognitive defect) which prevents understanding of, or adherence to the protocol
* Subject who in the opinion of the Investigator, require ACEi/ARB therapy post-transplant for any indication
* Subject who requires induction with Thymoglobulin, Campath, antithymocyte globulin (ATG), antilymphocyte globulin (ALG) or any biological induction agent other than basiliximab. Unplanned post-transplant use of these prohibited drugs for clinical indications post-transplant is allowed
* Subject has plans to become pregnant within 2 years post-transplant
* Subject who has a positive T-cell or B-cell crossmatch. Subjects with a weakly positive B-cell cross-match that tests negative following DTT reduction are acceptable
* Subject who has a requirement for maintenance immunosuppressant therapy with the exception of low dose steroid or mycophenolate mofetil (MMF). A subject who is on low dose tacrolimus maintenance therapy will be eligible provided the tacrolimus is withheld at least 1 week prior to transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2009-08-17 (Actual); Primary Completion 2015-05-11 (Actual); Study Completion 2018-04-03 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with the Presence of Allograft Interstitial Fibrosis and Tubular Atrophy (IF/TA) as Assessed at a Central Pathology Lab | up to 24 months
Progression of IF/TA from Month 6 to Month 24 | up to 24 months

SECONDARY OUTCOMES:
Time to T-cell Banff Mediated Rejection as Assessed at a Central Pathology Lab | up to 24 months
Percentage of Participants in Each Category of Banff 2007 Diagnostic Classification of Renal Allograft Pathology | up to 24 months
Percentage of Participants with Humoral Rejections | up to 24 months
Percentage of Participants with Acute Rejections | up to 24 months
Time to First Any Acute Rejection | up to 24 months
Banff 2007 Individual Sub-scores | up to 24 months
  Banff 2007 sub-scores (AH = Arteriolar hyalinethickening score; AT = Tubulitis score; AV = Intimal arteritis score; AI = Interstitial inflammation score; AG = Glomerulitis score; CG = Glomerulopathy score; CI = Interstitial fibrosis score; CT = Tubularatrophy score; CV = Vascular fibrous intimal thickening score; MM = Mesangial matrix increase score; TI = Total interstitial inflammation score; PTC = Peritubulary capillaritis score) is measured on an ordinal scale of 0 - 3.
Change from Baseline in Chronic Allograft Damage Index | Baseline and 6, 24 months
Percentage of Participants with Circulating Anti-Donor Antibody | up to 5 years
Number of Participants with Cellular Immune Response (ELISPOT) | up to 6 months
Urine Renal Biomarkers | up to 24 months
Graft Survival | up to 5 years
Patient Survival | up to 5 years
Renal Function as Measured by Glomerular Filtration Rate (GFR) | up to 5 years
Renal Function as Measured by Serum Creatinine | up to 5 years
Renal Function as Measured by Ratio of Urine Protein and Creatinine Concentrations | up to 5 years
12-Item Short Form (SF-12) Health Survey: Physical Composite Score (PCS) and Mental Health Composite Score (MCS) | up to 24 months
  The PCS and MCS are measured on a normalized 0-100 scale and computed using the corresponding subdomains from the SF-12 with 0 being the lowest level of health and 100 the highest.
Kidney Transplant Recipient Opinions of Immunosuppressive Medications Questionnaire | up to 24 months
  This questionnaire consists of 11 questions regarding immunosuppressive medications, where questions 1-3 ask about your experiences and opinions of transplant anti-rejection medications, questions 4 and 11 ask to rate each medication on the scale of 1-10, with 1 meaning disagree completely and 10 meaning agree completely, and questions 5-10 ask which medication satisfies the question.
Percentage of Participants with Polyomavirus Infection | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, Principal Investigator — University of Alberta; Use Central Contact, Study Director — Astellas Pharma Canada, Inc.
Locations (13):
- Canada (13):
  - Site CA133 Foothills Medical Centre, Calgary, Alberta
  - Site CA54 University of Alberta Hospital, Edmonton, Alberta
  - Site CA141 Health Sciences Centre, Winnipeg, Manitoba
  - Site CA114 Capital District Health Authority- QEII Health Sciences Centre, Halifax, Nova Scotia
  - Site CA150 St. Joseph's Healthcare, Hamilton, Ontario
  - Site CA27 London Health Sciences Centre, London, Ontario
  - Site CA165 St. Michael's Hospital, Toronto, Ontario
  - Site CA238 Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - Site CA172 Hôpital Notre-Dame du CHUM, Montreal, Quebec
  - Site CA144 McGill University Health Centre, Montreal, Quebec
  - Site CA64 Centre Hospitalier Universitaire de Québec- L'Hôtel-dieu de Québec, Québec, Quebec
  - Site CA116 Centre Hospitalier Universitaire de Sherbrooke- Hôpital Fleuirmont, Sherbrooke, Quebec
  - Site CA142 St. Paul's Hospital, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Campbell PM, Cantarovich M, Gangji A, Houde I, Jevnikar AM, Monroy-Cuadros FM, Nickerson PW, Paquet MR, Prasad GVR, Senecal L, Wolff JL, Schwartz JJ, Rush DN. A Five-Year Prospective, Randomized, Open-Label Study of Standard-Dose Versus Low-Dose Prolonged-Release Tacrolimus With or Without Angiotensin-Converting Enzyme Inhibitor or Angiotensin II Receptor Blocker Post Kidney Transplantation. Clin Transplant. 2025 Jan;39(1):e70067. doi: 10.1111/ctr.70067. PMID 39739990
- [Derived] Natale P, Mooi PK, Palmer SC, Cross NB, Cooper TE, Webster AC, Masson P, Craig JC, Strippoli GF. Antihypertensive treatment for kidney transplant recipients. Cochrane Database Syst Rev. 2024 Jul 31;7(7):CD003598. doi: 10.1002/14651858.CD003598.pub3. PMID 39082471
- [Derived] Cockfield SM, Wilson S, Campbell PM, Cantarovich M, Gangji A, Houde I, Jevnikar AM, Keough-Ryan TM, Monroy-Cuadros FM, Nickerson PW, Paquet MR, Ramesh Prasad GV, Senecal L, Shoker A, Wolff JL, Howell J, Schwartz JJ, Rush DN. Comparison of the effects of standard vs low-dose prolonged-release tacrolimus with or without ACEi/ARB on the histology and function of renal allografts. Am J Transplant. 2019 Jun;19(6):1730-1744. doi: 10.1111/ajt.15225. Epub 2019 Feb 1. PMID 30582281
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/hcp/study.aspx?ID=315